CLINICAL TRIAL: NCT06068556
Title: Safety, Reactogenicity and Immunogenicity Study of the Vector Vaccine GamCovidVac-M for the Prevention of Coronavirus (COVID-19) Infection Caused by the SARS-CoV-2 Virus With Altered Antigenic Composition With Participation of 12-17 Years Old Volunteers.
Brief Title: Study of the Vector Vaccine GamCovidVac-M (Altered Antigenic Composition)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13-GamCovidVac-M/N-2023
Record Dates: First submitted 2023-09-22; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy patients (Experimental): Drug: GamCovidVac-M vector vaccine for the prevention of COVID-19 with altered antigenic composition. A total of 50 people will be randomized and receive the study drug. Two intramuscular injections of GamCovidVac-M vector vaccine for the prevention of COVID-19 with altered antigenic composition will be performed. 1st injection - component I, 2nd injection - component II.
  Interventions: Biological: GamCovidVac-M vector vaccine for the prevention of COVID-19 with altered antigenic composition

INTERVENTIONS:
Biological: GamCovidVac-M vector vaccine for the prevention of COVID-19 with altered antigenic composition — Two intramuscular injections of GamCovidVac-M vector vaccine for the prevention of COVID-19 with altered antigenic composition will be performed. 1st injection - component I, 2nd injection - component II.

SUMMARY:
Safety, reactogenicity and immunogenicity study of the vector vaccine GamCovidVac-M for the prevention of coronavirus (COVID-19) infection caused by the SARS-CoV-2 virus with altered antigenic composition with participation of 12-17 years old volunteers.

ELIGIBILITY:
Inclusion Criteria:

The study will include volunteers who meet all the specified criteria:

1. Written informed consents to participate in the study, obtained from: the volunteer, his/her parent or a legal guardian;
2. 12-17 years old teenagers (men and women);
3. A negative test result for COVID-19, determined by PCR or express method before the introduction of the investigational medicinal product (IMP);
4. No COVID-19 during 6 months prior to the screening (according to the anamnesis);
5. No contact of the volunteer with COVID-19 patients for at least 14 days prior to inclusion in the Study (according to the volunteer, his/her parent or a legal guardian);
6. Consent to the use of effective methods of contraception during the entire period of participation in the Study;
7. A negative pregnancy test based on the results of a urine test at a screening visit (for women with preserved reproductive potential);
8. Negative test for the presence of narcotic and psychostimulants in the urine at the screening visit;

8. Negative alcohol content test at the screening visit; 9. No history of pronounced post-vaccination reactions or post-vaccination complications after the use of immunobiological drugs (according to the anamnesis); 9. Absence of acute infectious and/or respiratory diseases for at least 14 days prior to inclusion in the Study.

Exclusion Criteria:

Volunteers cannot be included in the study if there is at least one of the following criteria for non-inclusion:

1. Any vaccination/immunization carried out within 30 days prior to inclusion in the Study;
2. Therapy with steroids (with the exception of hormonal contraceptives and/or hormone replacement therapy) and / or immunoglobulins or other blood products that did not end 30 days before inclusion in the Study;
3. Therapy with any immunosuppressive drugs completed less than 3 months prior to inclusion in the Study;
4. Acute coronary syndrome or stroke suffered less than one year prior to inclusion in the Study;
5. Any immunodeficiency (for example, hereditary immunodeficiency, acquired immunodeficiency syndrome [AIDS], etc.);
6. Infectious diseases (according to the anamnesis): history of HIV, hepatitis, active form of syphilis at the time of screening; Tuberculosis; Active infection (with the exception of onychomycosis), or any acute infection episode requiring treatment with antibiotics intravenously for 4 weeks prior to screening or orally for 2 weeks prior to screening; History (according to the anamnesis) of serious recurrent or chronic infection, not listed above;
7. Extensive surgery within 4 weeks prior to screening;
8. Chronic autoimmune diseases or systemic collagenoses (according to the anamnesis), requiring the prescription of immunosuppressive therapy;
9. Volunteers who have undergone organ transplantation, including bone-marrow transplantation or peripheral blood stem cell transplantation and receive immunosuppressive therapy;
10. Splenectomy (according to the anamnesis);
11. Volunteers with a previous or concomitant history of neoplasms (ICD codes C00-D09);
12. Burdened allergic anamnesis (record of anaphylactic shock, Quincke's edema, polymorphic exudative eczema, serum sickness in the anamnesis), hypersensitivity or allergic reactions to the administration of immunobiological drugs, known allergic reactions to any of the components of the vaccine or vaccine containing similar components, exacerbation of allergic diseases on the day of inclusion in the study;
13. Neutropenia (decrease in the absolute number of neutrophils less than 1000 cells / mm3), agranulocytosis, significant blood loss, severe anemia (hemoglobin concentration less than 80 g/l), thrombocytopenia (decrease in the absolute number of platelets less than 50,000 cells/ mm3);
14. Anorexia, protein deficiency of any origin;
15. Volunteers with a BMI value in the range from -2 SD to +2 SD, according to their age;
16. Extensive tattoos at the injection sites (deltoid muscle area), which do not allow to assess the local reaction to the introduction of investigational medicinal product (IMP);
17. Chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, as well as diseases of the gastrointestinal tract, liver, kidneys, muscle and connective tissue in the stage of exacerbation or decompensation;
18. Presence of mental abnormalities (registered as psychiatrist's/narcologist's patient);
19. Diseases, the presence of which, from the point of view of the research doctor, puts the participant's health at risk in case of participation in the Study or potentially complicates the interpretation of the results of the examination;
20. Family members of the staff of research centers directly involved in the research;
21. The subject's participation in any other clinical trial 90 days prior to the screening;
22. Planned vaccination against COVID-19 with any vaccine, both in the framework of other studies and civil circulation;
23. Vaccination against COVID-19 or transmitted coronavirus infection COVID-19 less than 6 months prior to the screening;
24. Female volunteers during pregnancy or lactation;
25. Inability to read in Russian; inability or unwillingness to understand the essence of the Study. Any other conditions that limit the validity of obtaining informed consent or may affect the ability of a volunteer to participate in the Study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events (AE) | Within 7 days after each administration of the drug
  Occurrence of adverse events (AE)
Occurrence of serious adverse events (SAEs) | Through study completion, an average of 1 year
  Occurrence of serious adverse events (SAEs)

IPD SHARING:
Plan to Share IPD: Undecided